CLINICAL TRIAL: NCT06469684
Title: A Culturally-responsive Health Communication Intervention for Malay-Muslim Women on Breast Cancer Screening
Brief Title: A Health Education Intervention Tailored for Malay-Muslim Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Islamic Religious Council of Singapore (Unknown); National University Polyclinics, Singapore (Other)
Responsible Party: Principal Investigator, Wong Mee Lian, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NUS-IRB-2022-662
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Mammogram, Education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a matched pair cluster randomised controlled trial. Mosques in intervention and control arm are matched based on the region. Sessions within the same region (one intervention mosque and one control mosque) run parallel.
Who Masked: Participant
Masking Description: Randomisation done at mosque level. Allocation was not masked from individuals recruiting and delivering the interventions in the mosque.
  All participants within the same mosque receive the same intervention. Thus participants are only notified of the session conducted in the mosque they were recruited in.All participants are masked from the sessions conducted in other mosques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm receive health promotion intervention on breast cancer and mammogram including Mammobus deployment.
  Interventions: Behavioral: Health education session
- Control (Placebo Comparator): This arm receive health promotion intervention on healthy lifestyle.
  Interventions: Behavioral: Health education session

INTERVENTIONS:
Behavioral: Health education session — 1 hour health education session religious teaching promoting health-seeking behaviour, and question and answer session with healthcare professional.

SUMMARY:
The goal of this experimental study is to compare mammogram rate and knowledge in healthy women of Malay ethnicity in Singapore. The main questions it aims to answer are:

* Will health promotion intervention in the mosque on breast cancer and mammogram lead to mammogram uptake?
* Will health promotion intervention in the mosque on breast cancer and mammogram lead to change in knowledge and perception related to mammogram uptake? Participants will attend an education session in the mosque on breast cancer and mammogram by religious teacher and healthcare professional and will be given an opportunity to voluntarily sign up for mammogram on the Mammobus which will be deployed to the mosque.

Researchers will compare with healthy women of Malay ethnicity attending education session in the mosque on healthy lifestyle to see if there is a difference in mammogram uptake, and in knowledge and perception towards breast cancer and mammogram.

DETAILED DESCRIPTION:
The study will be a cluster randomized controlled trial of mosques to evaluate the impact of the education intervention. Each mosque is a cluster and intervention will be administered on a cluster level. We constructed a sampling frame of 29 large residential mosques out of the 70 mosques in Singapore. We excluded non-residential mosques and small mosques as these mosques do not conduct religious classes. From this sampling frame, we selected all 12 mosques that fulfilled the following eligibility criteria: i) a distance of at least 3.0 km from each other, to reduce bias of contamination, ii) availability of a parking space or an open area nearby for the MammoBus, and iii) high proportion of female mosque attendees as indicated by the Islamic Religious Council of Singapore (MUIS) which oversees the mosques in Singapore. We invited 12 mosques and received agreement from 6 mosques (clusters) for this trial. We stratified the mosques into 3 major housing estate regions (i.e. west, central and north), for stratified block randomization. Two mosques within each block or region were randomized by an independent researcher who is not on the study team, to the intervention arm and control arm (allocation ratio 1:1) using the ralloc package of STATA statistical software. Allocation will not be concealed. Three mosques on the intervention arm will receive the intervention package on breast cancer screening and three mosques on the control arm will receive an intervention package on healthy lifestyle. A total of 660 women will be recruited for the study by the research team on mosque grounds. All data collection is estimated to complete in 8 months.

Participants in the intervention arm will have three research visits and one optional research visit, therefore four research visits in total. Participants in the control arm will have three research visits in total. In both arms, all research visits will be conducted on mosque grounds. Mosque officers will allot time at the start or end of religious classes attended by potential participants to the research team to explain on the research study. Interested participants may approach interviewer in the mosque to sign up for the study. During recruitment, interviewer will go through the Participant Information Sheet and obtain verbal Informed Consent before conducting a baseline questionnaire. Only participants from the intervention arm will be asked for consent to be re-contacted for recruitment for a future study, a focus group discussion as the future study is not applicable for the control arm. Participant will be able to choose to attend one of the two available education sessions that will be held in the mosque over the next two weeks. Participant will be given a participant card to help them keep track of the dates of the session. The education session will be the second research visit for both arms. The third research visit is a voluntary session for those in the intervention arm, where participants may take part in a mammogram screening session in the mosque. The final research visit for both arms, fourth and third for intervention and control arm respectively, will take place between 2 months (± 1 month is applicable) from the recruitment, where a post-intervention survey will be carried out in the mosque. During this final research visit, participants that consented to be re-contacted for recruitment of a future follow-up study will be invited to participate in the follow-up study which is a focus group discussion.

Intervention package - i) Breast Cancer Screening: Participant will be required to complete a baseline questionnaire (10-15 minutes) upon recruitment and consent. Following recruitment, participant will be required to attend a group-level education session on breast cancer screening in the Malay language. This education session will last for an hour: 25 minutes education session by religious leaders on health-promoting Islamic teachings specifically on punitive religious beliefs, 10 minutes video on positive screening experience and breast cancer journey by breast cancer survivors, and 25 minutes question and answer on breast cancer by Malay-speaking health care provider. Participants will be asked to complete a short feedback form on the session. Participant will be given an educational pamphlet to reinforce health messages from the session and will be invited to attend a mammogram screening on the MammoBus. Participant may approach interviewers to sign up for the mammogram or register through the QR Code available on the participant card. This mammogram screening is voluntary and will be carried out in a MammoBus that will be deployed to the mosque in the following 2 weeks. The mammogram service is outsourced to National Healthcare Group Diagnostics (NHGD), that manages the MammoBus. The research team will only be involved in organising the mammogram appointments. Mammogram screening is a standard procedure in Singapore. In this research, mammogram screening will be according to the standard procedures and will be conducted by the trained radiographers from NHGD. Including waiting time and registration, this session should last for approximately 1 hour. Cost of mammogram screening will be borne by participants, where applicable. NHGD will inform participants of the results via mail when available. The research team and NUS as a whole will not have access to the mammogram results of the participants. At follow-up, 2 months (± 1 month is applicable) from the recruitment, participant will be required to answer a post-intervention questionnaire (10-15 minutes) which will be similar as the baseline survey, to measure changes in perception.

ii) Healthy lifestyle: Participant will be required to complete a baseline survey (10-15 minutes) upon recruitment and consent. Next, the participant will attend a group-level education session on healthy lifestyle in the Malay language. This education session will last for an hour - 30 minutes education session by religious leaders on health-promoting Islamic teachings, and 30 minutes question and answer on healthy lifestyle by Malay-speaking health care provider. Participants will be asked to complete a short feedback form on the session. At follow-up, 2 months (± 1 month is applicable) from the recruitment, participant will be required to answer a post-intervention questionnaire (10-15 minutes) which will be similar as the baseline questionnaire, to measure changes in perception.

Questionnaire and data collection - All data collected through questionnaires (pre-intervention questionnaire, feedback form and post-intervention questionnaire) will be linked via a unique code which will be given to the participant at recruitment and only this code will be used on all data. A separate encrypted file containing personal data of participants (i.e. phone number, name) linked to their unique code will be available only to the study administrator who is managing the service operations (i.e.arranging follow-up sessions and sending text reminders) of the study. A separate encrypted file containing personal data of participants that choose to go for mammogram (i.e. name, NRIC, phone number, address and date of birth) will be available only to the study administrator who is managing the mammogram appointments. Upon completion of all follow-up, recruitment for the follow-up study or completion of the mammogram appointment, whichever later, the files will be deleted therefore irreversibly de-identifying the data.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Malay-Muslim woman
* Aged 50-69
* Citizens or permanent residents of Singapore
* No history of breast cancer
* Had not gone for mammogram screening in the last 2 years

Exclusion Criteria:

* No basic fluency in the Malay language
* Not able to provide a coherent response
* Declined photography of the education session

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence Rate Ratio of Mammogram Uptake by Arm | 2-3 months
  Attending mammogram after health education session

SECONDARY OUTCOMES:
Incidence Rate Ratio of Knowledge and Perception at Follow-up by Arm, adjusting for baseline | 2-3 months
  Survey output on knowledge and perception on health behaviour, breast cancer and mammogram

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
De-identified survey data will be shared only upon request due to privacy and ethical concerns